CLINICAL TRIAL: NCT03967665
Title: Risk Stratification-directed N-acetyl-L-cysteine for Prevention of Poor Hematopoietic Reconstitution After Unmanipulated Haploidentical Stem Cell Transplantation--an Open-label, Randomized, Controlled, Clinical Trial
Brief Title: Risk Stratification-directed NAC for Prevention of Poor Hematopoietic Reconstitution
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Supervisor of Hematology,Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NAC prevention of PGF and PT
Record Dates: First submitted 2019-04-03; First posted 2019-05-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Stem Cell Transplant Complications
Keywords: N-acetyl-L-cysteine; Poor hematopoietic reconstitution; Unmanipulated Haploidentical stem cell Transplantation
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): NAC 400 mg three times per day from -14D pre-HSCT to +2 months
  Interventions: Drug: N-acetyl-L-cysteine
- Control arm (No Intervention): No-NAC concurrent control according to a 2:1 schedule.

INTERVENTIONS:
Drug: N-acetyl-L-cysteine — NAC 400 mg three times per day from -14D pre-HSCT to +2 months post-HSCT
  Other Names: NAC
  Arms: Treatment arm

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment of malignant hematopoietic diseases. However, poor hematopoietic reconstitution including poor graft function (PGF) and prolonged isolated thrombocytopenia (PT), remains a life-threatening complication after allo-HSCT. Especially with the increasing use of haploidentical allo-HSCT (haplo-HSCT) in the past ten years, PGF and PT have become growing obstacles contributing to high morbidity and mortality after allo-HSCT. Due to the limited mechanism studies, the clinical management of PGF and PT is challenging.

Recent prospective case-control studies reported that the reduced and dysfunctional bone marrow (BM) endothelial cells (ECs) after allo-HSCT are involved in the pathogenesis of PGF and PT. Moreover, in vitro treatment with N-acetyl-L-cysteine (NAC) could enhance the defective hematopoietic stem cell (HSC) function through repairing the dysfunctional BM ECs of PGF and PT patients. The investigators performed a small-scale pilot cohort study and saw encouraging clinical results that oral administration with NAC could partially repair the dysfunctional BM ECs and improve megakaryocytopoiesis in PT patients, which suggests that NAC is a promising drug in PT patients after allo-HSCT. In addition, prior prospective trial of the investigators suggests that BM ECs<0.1% pre-HSCT is the risk factor for occurrence of the PGF and PT two months following allo-HSCT. Previous single-arm clinical cohort studies of the investigators showed that prophylactic use of NAC before allo-HSCT reduced the incidence of poor hematopoietic reconstitution after allo-HSCT in patients with ECs <0.1% pre-HSCT.

Therefore, the investigators designed the study with acute leukemia patients who will be scheduled to receive haplo-HSCT. The patients who are in the first complete remission at time of haplo-transplant will be enrolled in the study. Exclusive criteria are bronchila asthma and NAC allergy. The enrolled patients were risk-stratified into BM ECs≥0.1% group (low-risk group) and BM ECs<0.1% group (high-risk group). Patients in high-risk group (ECs<0.1%) will be randomized to 1 of 2 arms: (a) NAC 400 mg three times per day from 14 days pre-HSCT to 2 months post-HSCT, (b) No-NAC concurrent control according to a 2:1 schedule. The aim of the trail is to assess the effects of NAC for prevention of poor hematopoietic reconstitution in patients with acute leukemia undergoing haplo-HSCT.

DETAILED DESCRIPTION:
This study is designed as a phase III, open-label, randomized study assessing the safety and efficacy of NAC (400 mg, orally, three times daily) versus no-NAC control for prevention of poor hematopoietic reconstitution in patients with acute leukemia undergoing haploidentical HSCT in a 2:1 ratio. The study will consist of three phases: a pre-randomization phase, a treatment phase, and an observational follow-up phase.

The screening period: Patients will be screened during a 1 week screening period prior to entering the trial to allow for the collection of BM samples to evaluate the quantity and function of BM ECs at 21-14 days before HSCT. The enrolled patients were risk-stratified into BM ECs≥0.1% group (low-risk group) and BM ECs<0.1% group (high-risk group). Approximately 126 patients with BM EC <0.1% at day-14 pre-HSCT (84 patients in NAC treatment arm and 42 patients in control arm) will be randomized in a 2:1 ratio to 1 of 2 arms: (a) NAC 400 mg three times per day, (b) No-NAC concurrent control.

The treatment phase: Study medication will be administered orally, 400 mg three times daily from -14 days pre-HSCT to +2 months post-HSCT. All patients should continue their pre study dose of NAC throughout trial participation. Following randomization, patients will have 3 hospitalized or at-clinic trial visits at day 0 before-HSCT and 1, 2 months post-HSCT to evaluate efficacy, safety, tolerability and compliance with study medication. Patients will be contacted by trial site staff on a monthly basis between visits beginning with day 0.

The observational follow-up phase: Upon completion of the trial participation phase all eligible patients will enter an open label follow-up phase. Clinic visits will occur every 3 months (± 1 week).

Patients will have a pretreatment bone marrow aspiration conducted and have a follow up bone marrow aspiration conducted at day0 before-HSCT and 1, and 2 months post-HSCT. All patients who complete or discontinue from the trial, for any reason, will have a follow up visit, 4 weeks after their last dose of study medication. The primary outcome is the incidence of PGF and PT at 2 months after HSCT, as well as the safety. Secondary endpoints included cumulative incidences of relapse (CIR), acute graft-versus-host disease (aGVHD), non-relapse mortality (NRM), overall survival (OS), disease free survival (DFS), the related laboratory evaluation of ECs and HSC in BM microenvironment, etc.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia in the first complete remission (CR1) at time of haplo- transplant.
* Age ≥ 15 years.
* Contraception: Female patients of childbearing potential must use ≥ 1 effective (≤ 1% failure rate) method of contraception during the trial and until the end of treatment visit.
* Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

* History or presence of allergy to NAC.
* History or presence of clinically concerning Bronchial asthma.
* Non-CR1 leukemia at time of transplant.
* Patients undergoing transplant from donors other than haploidentical relatives.
* Patients who have previously participated in a clinical trial of NAC.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of poor hematopoietic reconstitution at 2 months post-HSCT | 2 months post-HSCT
  The incidence of poor hematopoietic reconstitutio at 2 months post-HSCT

SECONDARY OUTCOMES:
Cumulative incidences of relapse at one year post-HSCT | 1 year after transplantation
  Cumulative incidences of relapse at one year post-HSCT.
Cumulative incidences of acute graft-versus-host disease for 100 days post-HSCT | 100 days after transplantation
  Cumulative incidences of acute graft-versus-host disease for 100 days post-HSCT
Non-relapse mortality during 1 year post-HSCT | 1 year after transplantation
  Non-relapse mortality during 1 year post-HSCT
Overall survival during 1 year post-HSCT | 1 year after transplantation
  Overall survival during 1 year post-HSCT
Disease free survival during 1 year post-HSCT | 1 year after transplantation
  Disease free survival during 1 year post-HSCT
Number of participants with treatment-related adverse events during oral administration of NAC. | 14 days pre-HSCT to 2 months post-HSCT.
  Number of participants with treatment-related adverse events during oral administration of NAC.
Effect of NAC on ECs percentage at 0 day pre-HSCT, 1 month, 2 months post-HSCT | 0 day pre-HSCT, 1 month, 2 months post-HSCT
  ECs percentages at 0 day pre-HSCT, 1 month, 2 months post-HSCT
Effect of NAC on HSCs percentagesat 0 day pre-HSCT, 1 month, 2 months post-HSCT | 0 day pre-HSCT, 1 month, 2 months post-HSCT
  HSCs percentages at 0 day pre-HSCT, 1 month, 2 months post-HSCT
Effect of NAC on MKs numbers at 0 day pre-HSCT, 1 month, 2 months post-HSCT | 0 day pre-HSCT, 1 month, 2 months post-HSCT
  MKs numbers at 0 day pre-HSCT, 1 month, 2 months post-HSCT
Incidence of viral infection until 100 days post-HSCT. | 100 days post-HSCT.
  Incidence of viral infection until 100 days post-HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Kong Y, Zhao HY, Zhang YY, Wang YZ, Xu LP, Zhang XH, Liu KY, Huang XJ. Prophylactic NAC promoted hematopoietic reconstitution by improving endothelial cells after haploidentical HSCT: a phase 3, open-label randomized trial. BMC Med. 2022 Apr 27;20(1):140. doi: 10.1186/s12916-022-02338-9. PMID 35473809